CLINICAL TRIAL: NCT06561022
Title: Precision Treatment of HR+ HER2- Advanced Breast Cancer Based on SNF Molecular Subtyping
Acronym: abemaSNF1/3
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N038
Record Dates: First submitted 2024-07-21; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
Keywords: abemeciclib; subtyping -based medicine; post-CDK4/6 inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — fluzoparib; Everolimus; Fulvestrant; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SNF 1 safety lead-in phase (Experimental): Everolimus plus Fulvestrant and Abemaciclib in patients with HR+ HER2-advanced breast cancer of SNF1 subtype who have progressed after CDK4/6 inhibitor treatment.
  Interventions: Drug: Everolimus; Drug: Fulvestrant; Drug: Abemaciclib
- SNF 1 Phase II Control (Active Comparator): Fulvestrant and Abemaciclib in patients with HR+ HER2-advanced breast cancer of SNF1 subtype who have progressed after CDK4/6 inhibitor treatment.
  Interventions: Drug: Fulvestrant; Drug: Abemaciclib
- SNF 1 Phase II Experimental (Experimental): Everolimus plus Fulvestrant and Abemaciclib in patients with HR+ HER2-advanced breast cancer of SNF1 subtype who have progressed after CDK4/6 inhibitor treatment.
  Interventions: Drug: Everolimus; Drug: Fulvestrant; Drug: Abemaciclib
- SNF 3 safety lead-in phase (Experimental): Fluzoparib plus Fulvestrant and Abemaciclib in patients with HR+ HER2-advanced breast cancer of SNF3 subtype who have progressed after CDK4/6 inhibitor treatment.
  Interventions: Drug: Fluzoparib; Drug: Fulvestrant; Drug: Abemaciclib
- SNF 3 Phase II Control (Active Comparator): Fulvestrant and Abemaciclib in patients with HR+ HER2-advanced breast cancer of SNF3 subtype who have progressed after CDK4/6 inhibitor treatment.
  Interventions: Drug: Fulvestrant; Drug: Abemaciclib
- SNF 3 Phase II Experimental (Active Comparator): Fluzoparib plus Fulvestrant and Abemaciclib in patients with HR+ HER2-advanced breast cancer of SNF3 subtype who have progressed after CDK4/6 inhibitor treatment.
  Interventions: Drug: Fluzoparib; Drug: Fulvestrant; Drug: Abemaciclib

INTERVENTIONS:
Drug: Fluzoparib — Fluzoparib
  Arms: SNF 3 Phase II Experimental; SNF 3 safety lead-in phase
Drug: Everolimus — Everolimus
  Arms: SNF 1 Phase II Experimental; SNF 1 safety lead-in phase
Drug: Fulvestrant — Fulvestrant
Drug: Abemaciclib — Abemaciclib

SUMMARY:
To explore the efficacy and safety of Everolimus (SNF1 subtype) or Fluzoparib (SNF3 subtype) combined with Fulvestrant and Abemaciclib vs. Fulvestrant combined with Abemaciclib in patients with HR+/HER2- breast cancer of SNF1/SNF3 subtype who have progressed after CDK 4/6 inhibitor treatment.

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label, phase II study to explore the efficacy and safety of a three-drug combination of Everolimus or Fluzoparib plus Fulvestrant and Abemaciclib compared to a two-drug combination of Fulvestrant plus Abemaciclib in patients with HR+ HER2-advanced breast cancer of SNF1/SNF3 subtype who have progressed after CDK 4/6 inhibitor treatment. The study consists of Safety Lead-in phase, which aims to explore the safety and preliminary efficacy of the three-drug combination, and phase II, which aims to explore the efficacy of the three-drug combination.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be enrolled in this study:

  1. Females aged ≥ 18 years and ≤ 70 years.
  2. Histologically confirmed HR-positive HER2-negative (specific definition: tumors are defined as ER positive when ≥ 1% tumor cells are positive by immunohistochemistry (IHC), and tumors are defined as HER2 negative when HER2 is 0-1+ or HER2 is ++ but the FISH or CISH result is negative and no amplification) locally advanced breast cancer (no radical local treatment is possible) or recurrent metastatic breast cancer with digital pathological staging of SNF1 or SNF3 subtype.
  3. Progression after CDK 4/6 inhibitor treatment. If CDK 4/6 inhibitors are used in the adjuvant treatment, metastatic relapse should occur during the administration of CDK 4/6 inhibitor or within 12 months after the end of the administration. If CDK 4/6 inhibitors are used in the first-line treatment for metastatic relapse, disease progression should occur during the administration.
  4. Have received ≤ first-line systemic therapy after metastatic relapse.
  5. Have at least one assessable lesion according to RECIST version 1.1.
  6. The patient has adequate organ function for all of the following criteria, as defined below:

     Hematologic: HB ≥ 90 g/L (no transfusion within 14 days); ANC ≥ 1.5 × 109 /L; PLT ≥ 100 × 109 /L.
  7. Hepatic: TBIL ≤ 1.5 × ULN (upper limit of normal) Patients with Gilbert's syndrome with a total bilirubin ≤ 2.0 times ULN and direct bilirubin within normal limits are permitted. ALT and AST ≤ 3 × ULN; serum Cr ≤ 1 × ULN, endogenous creatinine clearance > 50 mL/min (Cockcroft-Gault formula).
  8. Have not received endocrine therapy, targeted therapy, and surgery within 3 weeks prior to the start of the study and have recovered from acute toxic reactions to previous treatment (if surgery was performed, the wound has fully healed).
  9. Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and randomization.
  10. Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to randomization. A washout period of at least 21 days is required between last chemotherapy dose and randomization (provided the patient did not receive radiotherapy).
  11. The patient is able to swallow oral medications.
  12. ECOG score ≤ 1 and life expectancy ≥ 3 months.
  13. Female subjects of childbearing potential are required to use a medically approved contraceptive measure during the study treatment and for at least 3 months after the last dose of investigational drug.
  14. Subjects are voluntarily enrolled in this study, have signed informed consent form, have good compliance and cooperate with follow-up.

Exclusion Criteria:

* Patients with any of the following could not be enrolled in this study:

  1. Use of radiotherapy within 3 weeks prior to treatment.
  2. Patients with known CNS metastases or a history of CNS metastases prior to screening. For patients with clinically suspected CNS metastases, enhanced CT or enhanced magnetic resonance imaging (MRI) must be performed within 28 days prior to the first dose to rule out CNS metastases.
  3. The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
  4. The patient has active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
  5. The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
  6. ≥ grade 1 adverse reactions due to previous treatment that are still ongoing. Exceptions are alopecia or the cases that, in the opinion of the investigator, should not be excluded. Such cases should be clearly documented in the investigator's notes.
  7. The patient has had major surgery within 14 days prior to randomization.
  8. Females who are pregnant or lactating.
  9. Malignant tumor within the past five years (except cured basal-cell carcinoma and cervical carcinoma in situ)
  10. Inability to swallow, chronic diarrhoea and intestinal obstruction, and the presence of multiple factors that affect the administration and absorption of medication.
  11. Presence of third spacing that cannot be controlled by drainage or other methods (e.g., large amounts of pleural effusion and ascites).
  12. Non-healing wounds for a long time or fractures that are not fully healed.
  13. Allergic individuals, or those with a known history of allergy to the components of the drug involved in this protocol.
  14. Long-term use of oral steroid hormones. For occasional use in the past, a 4-week discontinuation period is required before enrollment.
  15. Previous use of PAM pathway inhibitors such as Everolimus and PARP inhibitors such as Fluzoparib.
  16. Use of any chemotherapy drugs during metastatic relapse.
  17. Have received specific regimen of Abemaciclib combined with Fulvestrant during metastatic relapse (i.e., the control group in this study).
  18. Have received CDK 4/6 inhibitors for > 1 treatment period.
  19. The patient has received an experimental treatment in a clinical trial within the last 30 days or 5 half-lives, whichever is longer, prior to randomization, or is currently enrolled in any other type of medical research (for example: medical device) judged by the sponsor not to be scientifically or medically compatible with this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-08-21 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0( Safety lead-in Phase) | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
objective response rate (ORR)( Safety lead-in Phase) | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
  objective response rate (ORR)
Progression-free survival (PFS)(Phase II) | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
  Progression-free survival (PFS)

SECONDARY OUTCOMES:
Overall survival (OS)(Phase II) | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
  Overall survival (OS)
objective response rate (ORR)(Phase II) | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
  objective response rate (ORR)
clinical benefit rate (CBR)(Phase II) | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
  clinical benefit rate (CBR)
duration of response (DOR)(Phase II) | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
  duration of response (DOR)
time to first response (TTR)(Phase II) | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
  time to first response (TTR)
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0(Phase II) | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Clinical benefit rate (CBR)( Safety lead-in Phase) | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
  Clinical benefit rate (CBR)
Progression-free survival (PFS)( Safety lead-in Phase) | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
  Progression-free survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin C Shao, MD, PhD, Principal Investigator — Fudan U
Locations (1):
- 270 Dongan Road, Fudan University Shanghai Cancer Center, Shanghai, China